CLINICAL TRIAL: NCT00902616
Title: L-Arginine and Endothelial Dysfunction in Type 2 Diabetic Patients
Brief Title: Effect of Arginine on Microcirculation in Patients With Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tameside Hospital NHS Foundation Trust (Other)
Responsible Party: Mr Philip Dylak, Tameside General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Arginine01
Record Dates: First submitted 2009-05-12; First posted 2009-05-15 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2009-05

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Peripheral neuropathy; Microcirculation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Peripheral Nervous System Diseases | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. L-arginine (Active Comparator): 3 gm TDS for 3 months
  Interventions: Dietary Supplement: L-arginine
- 2. Placebo - Lactose powder (Placebo Comparator): 3 gm TDS for 3 months
  Interventions: Dietary Supplement: Placebo Lactose powder

INTERVENTIONS:
Dietary Supplement: L-arginine — 3gm TDS for three months
  Arms: 1. L-arginine
Dietary Supplement: Placebo Lactose powder — 3gm TDS for 3 months
  Arms: 2. Placebo - Lactose powder

SUMMARY:
Patients with diabetes have dysfunction of the lining of the arteries which lead to impaired circulation in the small blood vessels. This is thought to be secondary to reduced chemicals in the blood viz: nitric oxide. This chemical is derived from an amino acid (protein) L-arginine. Therefore, the researchers investigated whether giving patients L-arginine (versus dummy powder) would improve the blood flow in the small blood vessels in the lower limbs of patients with damage to their nerves (neuropathy).

DETAILED DESCRIPTION:
Peripheral neuropathy is one of the most common complications of diabetes mellitus (DM) with a prevalence of around 30 - 45%. In addition, diabetic patients are at increased risk of macrovascular disease, as well as other complications such as retinopathy and nephropathy.

The majority of patients will have developed peripheral neuropathy 10-20 years after the onset of diabetes, which is an important cause of foot ulceration, Charcot joints, amputation and increased morbidity and mortality. In view of this the cost to the National Health Service in 1987 was a staggering £13.5 million. Therefore there is an urgent need for prevention of diabetic neuropathy and its sequelae.

The exact pathogenesis of diabetic neuropathy is unclear, with both metabolic and vascular factors having been implicated. Microvascular disease is possibly the initial event in the development of diabetic complications. Microvascular disease may play an important role in the causation and exacerbation of diabetic neuropathy. Histopathological studies have shown thickening of vessel walls, hyperplasia of capillary endothelial cells and increased plugging of vessels in neuropathic patients. Endothelial dysfunction is thought to be an important initiating factor for the development of these complications. Endothelial dysfunction is thought to develop as a consequence of changes in nitric oxide and cell adhesion molecules in the plasma of diabetic patients. L-arginine is an amino acid, which is the only source of NO in the body.

We therefore propose to study the efficacy of arginine supplementation ( this is available over the counter as a food supplement) on endothelial function and other biomarkers of impaired endothelial function. We hope with this study to demonstrate that L-arginine supplementation will enhance nitric oxide availability, thereby improve the microcirculation and subsequently improve peripheral nerve function. We will use surrogate markers to assess the efficacy of L-arginine supplementation to show an improvement in diabetic complications such as microalbuminuria in the urine, and TcPO2 in the skin of the lower limbs. In addition microcirculation will be assessed using the Moor Laser Doppler flow machine and the Radiometer TcPO2 device. Endothelial function will also be assessed indirectly by measuring the cell adhesion molecules ICAM-1, VCAM-1, P-selectin and E-selectin. This will be performed using standard ELISA techniques.

A total of 40 patients will be recruited for the study. Half will be randomised to taking the food supplement L-arginine and half to placebo. At baseline all patient will have a clinical assessment of their neuropathy status in the lower limb, blood pressure and BMI. Fasting bloods for glucose, lipids profile, U&E's, FBC, CRP, cell adhesion molecules and nitric oxide will be done at baseline and three months later at the end of the study. The TcPO2 and micro-circulation will be assessed at baseline and also at three month.

Each of the twenty patients that is randomised to L-arginine will be given a tin containing 1 kilogram of the food supplement L-arginine. They are to take a spoonful (three grams) of the L-arginine and dissolve it in a glass of sugar free cold drink of their choice such as orange or lemon squash. They are to take it before food three times a day. The twenty patient randomised to placebo will receive a tin containing one kilogram of placebo and the instruction is as for the L-arginine group.

20 patients will receive L-arginine powder (3G TDS) and 20 patients will receive placebo, lactose powder (3G TDS)

Clinical examination as part of routine care:

1. BMI, BMI will be calculated by weight/height (kg/m2).
2. Lying and standing blood pressure will be measured twice, in the right arm using Dinamap™ (Critikon, UK), after resting for 10 minutes. Hypertension will be defined according to WHO criteria (systolic blood pressure (sBP) >140 mm Hg and/or diastolic blood pressure (dBP) >90 mm Hg or if the patient is on current antihypertensive treatment.
3. Overnight microalbumin excretion rate.
4. Neuropathic Disability Score and Vibration Perception threshold.

Additional examination:

1. TcPO2 of the right foot.
2. Micro-circulation of the right foot using Moore Laser Doppler iontophoresis.

Blood from an antecubital vein will be collected after an overnight fast and after resting for fifteen minutes in the supine position for:

1. as part of routine care - FBC, U&E's, fasting glucose, glycated haemoglobin, fasting lipid profile
2. additional blood test - CRP, cell adhesion molecules, nitric oxide

ELIGIBILITY:
Inclusion Criteria:

* Males and females diabetic patients with peripheral neuropathy, aged 30-65 years
* Type 2 diabetes (NIDDM) judged by WHO criteria:

  * onset of diabetes mellitus after the age of 30 years
  * not requiring insulin for control of diabetes or insulin treatment initiated after one year diagnosis of diabetes
  * no history of diabetic ketoacidosis
* All patients will have detailed history and physical examination

Exclusion Criteria:

* Patients with ischaemic heart disease
* Previous stroke and severe peripheral vascular disease)
* Previous amputation
* Renal failure (defined as serum creatinine > 120 mmol/l)
* Uncontrolled hypertension (BP > 160/90)
* Patients on nitrates

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2003-06; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Improvement in microcirculation | 3 months

SECONDARY OUTCOMES:
Effect of L-arginine on clinical parameters of neuropathy | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Edward Jude, MD, MRCP, Principal Investigator — Tameside General Hospital
Locations (1):
- Tameside General Hospital, Ashton-under-Lyne, Cheshire, United Kingdom